CLINICAL TRIAL: NCT00237523
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of IoGen™ for the Treatment of Moderate or Severe, Periodic Breast Pain Associated With Symptomatic Fibrocystic Breast Disease
Brief Title: Study for Treatment of Moderate or Severe, Periodic, "Cyclic", Breast Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Symbollon Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SYM1210
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-06

CONDITIONS: Fibrocystic Disease of Breast; Fibrocystic Changes of Breast; Fibrocystic Mastopathy; Pain
Keywords: Breast pain; Mastalgia; Cyclic mastalgia; Periodic mastalgia; Non-cyclic mastalgia; Fibrosis; Nodularity; Cysts; Fibrocystic breast disease; Fibrocystic breast condition; Fibocystic breast syndrome
MeSH Terms: conditions — Fibrocystic Breast Disease; Pain; Mastodynia; Fibrosis; Cysts | interventions — Iodides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IoGen (molecular iodine)

SUMMARY:
* History of clinical breast pain for at least the last six months.
* At least six days of moderate or severe breast pain per cycle.
* Fibrosis, cysts, nodules involving at least 25% of the surface of one breast.
* Euthyroid with no prior history of thyroid disease.
* Six months of daily therapy with molecular iodine.
* Placebo controlled vs active (1:1).

DETAILED DESCRIPTION:
Primary efficacy parameters will be measured by patient self-assessment of pain/tenderness using a categorical daily pain diary. Clinical pain is defined as a patient assessment of moderate or severe pain for any given day. Total clinical pain per menstrual cycle is calculated based upon the categorical ratings recorded in a patient's daily pain diary over the course of a complete menstrual cycle.

A directed breast examination will be used as a secondary efficacy endpoint. Changes in the brest examination will be determined by the physician after consideration of both the nature of the examination findings and the surface area of breast involvement. Changes as noted after six months of therapy, relative to the screening visit (baseline) will be used to evaluate this endpoint.

ELIGIBILITY:
Inclusion Criteria:

* History of clinical breast pain.
* Documentation of 6 or more sequential days of moderate or severe pain by patient daily diary.
* Conservative measures such as local heat, non-prescription analgesics, and properly fitted garments are not effective for the treatment of symptoms
* Euthyroid with no prior history of thyroid disease.
* Premenopausal female between the ages of 18 and 50.
* The presence of at least one palpable structure (nodules, cysts) and involvement (diffuse nodularity or breast thickening) of at least 25% of at least one breast surface.

Exclusion Criteria:

* History of thyroid disease
* Non-cyclic breast pain
* Treatment with gonadotropin releasing hormone (GnRH) agonist, Danocrine, tamoxifen, raloxifene, or bromocriptine within three months of starting the trial
* Initiation or change of any hormonal therapy within 6 months of enrollment; including birth control pills, hormone replacement therapy, any progestin including Norplant or Depo-Provera;
* Current treatment with iodine or iodine-containing medications or diagnostics
* Known hypersensitivity to iodine-containing products
* Breast implants;
* Oophorectomy (complete or partial)
* Uncontrolled hypertension;
* Breast biopsy breast biopsy within two months of screening; or expectation of a breast biopsy during the study for a suspicious mass present at baseline;
* Pregnant women or nursing mothers
* History of malignancy within the previous 5 years other than basal cell or squamous cell carcinoma of the skin
* History of breast cancer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 2005-07; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Total clinical breast pain as documented by patient daily diary.

SECONDARY OUTCOMES:
Change in fibrosis based upon breast examination.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kazakhin, M.D., Study Director — Symbollon Pharmaceuticals, Inc.
Locations (39):
- United States (39):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - Downtown Women's Heath Care, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - S.H.E. Medical Associates, Hartford, Connecticut
  - The GYN's Center for Women's Health, Waterbury, Connecticut
  - Greater Hartford Women's Health Associates, West Hartford, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Miami Research Associates, Inc., Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Physicians Research Group, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Kentucky Medical Research Center, Lexington, Kentucky
  - York Clinical Consulting, Marrero, Louisiana
  - MedVadis Research, Wellesley, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - University of Missouri, Kansas City, Missouri
  - Department of Ob/Gyn - Women's Health University of Saint Louis, St Louis, Missouri
  - The Medical Group of Northern Nevada, Reno, Nevada
  - Women's Health Research Center, LLC, Lawrenceville, New Jersey
  - Laurel Creek Research Associates, Moorestown, New Jersey
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - HWC Women's Research Center, Miamisburg, Ohio
  - LION Research, Norman, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Fellows Research Alliance, Inc., Hilton Head Island, South Carolina
  - Women's Clinical Research Center/North Seattle Women's Group, Seattle, Washington
  - Tacoma Women's Specialists, Tacoma, Washington

REFERENCES:
- [Background] Aceves C, Anguiano B, Delgado G. Is iodine a gatekeeper of the integrity of the mammary gland? J Mammary Gland Biol Neoplasia. 2005 Apr;10(2):189-96. doi: 10.1007/s10911-005-5401-5. PMID 16025225
- [Background] Cann SA, van Netten JP, van Netten C. Hypothesis: iodine, selenium and the development of breast cancer. Cancer Causes Control. 2000 Feb;11(2):121-7. doi: 10.1023/a:1008925301459. PMID 10710195
- [Background] Kessler JH. The effect of supraphysiologic levels of iodine on patients with cyclic mastalgia. Breast J. 2004 Jul-Aug;10(4):328-36. doi: 10.1111/j.1075-122X.2004.21341.x. PMID 15239792
- [Background] Ghent WR, Eskin BA, Low DA, Hill LP. Iodine replacement in fibrocystic disease of the breast. Can J Surg. 1993 Oct;36(5):453-60. PMID 8221402
- [Background] Garcia-Solis P, Alfaro Y, Anguiano B, Delgado G, Guzman RC, Nandi S, Diaz-Munoz M, Vazquez-Martinez O, Aceves C. Inhibition of N-methyl-N-nitrosourea-induced mammary carcinogenesis by molecular iodine (I2) but not by iodide (I-) treatment Evidence that I2 prevents cancer promotion. Mol Cell Endocrinol. 2005 May 31;236(1-2):49-57. doi: 10.1016/j.mce.2005.03.001. Epub 2005 Apr 13. PMID 15922087
- [Background] Eskin BA, Grotkowski CE, Connolly CP, Ghent WR. Different tissue responses for iodine and iodide in rat thyroid and mammary glands. Biol Trace Elem Res. 1995 Jul;49(1):9-19. doi: 10.1007/BF02788999. PMID 7577324
- [Background] Thrall KD, Bull RJ, Sauer RL. Distribution of iodine into blood components of the Sprague-Dawley rat differs with the chemical form administered. J Toxicol Environ Health. 1992 Nov;37(3):443-9. doi: 10.1080/15287399209531682. PMID 1433379
- [Background] Venturi S. Is there a role for iodine in breast diseases? Breast. 2001 Oct;10(5):379-82. doi: 10.1054/brst.2000.0267. PMID 14965610
- [Background] Smyth PP. Role of iodine in antioxidant defence in thyroid and breast disease. Biofactors. 2003;19(3-4):121-30. doi: 10.1002/biof.5520190304. PMID 14757962
- [Background] Ader DN, South-Paul J, Adera T, Deuster PA. Cyclical mastalgia: prevalence and associated health and behavioral factors. J Psychosom Obstet Gynaecol. 2001 Jun;22(2):71-6. doi: 10.3109/01674820109049956. PMID 11446156
- [Background] Ader DN, Shriver CD, Browne MW. Cyclical mastalgia: premenstrual syndrome or recurrent pain disorder? J Psychosom Obstet Gynaecol. 1999 Dec;20(4):198-202. doi: 10.3109/01674829909075596. PMID 10656154
- [Background] Ader DN, Browne MW. Prevalence and impact of cyclic mastalgia in a United States clinic-based sample. Am J Obstet Gynecol. 1997 Jul;177(1):126-32. doi: 10.1016/s0002-9378(97)70450-2. PMID 9240595